CLINICAL TRIAL: NCT02498600
Title: Phase II Randomized Trial of Nivolumab With or Without Ipilimumab in Patients With Persistent or Recurrent Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: Nivolumab With or Without Ipilimumab in Treating Patients With Persistent or Recurrent Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02424; NCI-2014-02424 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY003; 9698; NRG-GY003 (Other: NRG Oncology); NRG-GY003 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2015-07-14; First posted 2015-07-15 (Estimated); Results first posted 2020-09-11 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
Keywords: Phase II Randomized Trial of Nivolumab with or without Ipilimumab in Patients with Persistent or Recurrent Epithelial Ovarian; Primary Peritoneal or Fallopian; Tube Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (nivolumab) (Active Comparator): INDUCTION: Patients receive nivolumab IV over 30 minutes every 2 weeks. Treatment repeats every 4 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive nivolumab IV over 30 minutes every 2 weeks. Treatment repeats every 4 weeks for up to 21 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab
- Group II (nivolumab, ipilimumab) (Experimental): INDUCTION: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 90 minutes. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive nivolumab IV over 30 minutes every 2 weeks. Treatment repeats every 4 weeks for up to 21 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Group II (nivolumab, ipilimumab)
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This randomized phase II trial studies how well nivolumab works with or without ipilimumab in treating patients with epithelial ovarian, primary peritoneal, or fallopian tube cancer that has not responded after prior treatment (persistent) or has come back (recurrent). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the proportion of patients who have objective tumor response (complete or partial) by modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in patients with persistent or recurrent epithelial ovarian, fallopian tube, primary peritoneal cancers, treated with nivolumab or the combination of nivolumab and ipilimumab and to assess the difference in objective response rate (ORR) between patients treated with nivolumab versus those treated with the combination of nivolumab and ipilimumab.

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) hazard ratio for patients treated with nivolumab versus those treated with the combination of nivolumab and ipilimumab.

II. To estimate and compare the duration of overall survival (OS) for patients treated with nivolumab or the combination of nivolumab and ipilimumab.

III. To determine the frequency and severity of adverse events associated with treatment with nivolumab or the combination of nivolumab and ipilimumab as assessed by Common Terminology Criteria for Adverse Events (CTCAE).

IV. To determine whether cellular and molecular laboratory parameters in pre-treatment tissue and peripheral blood specimens predict overall survival (OS), tumor response by modified RECIST 1.1, and progression-free survival (PFS):

IVa. PD-L1 expression in tumor cells and tumor-infiltrating lymphocytes (TILs) measured by quantitative immunohistochemistry (IHC).

IVb. Natural anti-tumor immunity in tumor cells and TILs measured using IHC and T cell repertoire analyses.

IVc. Tumor "immunogenicity" as determined by the neo-epitope landscape using next-generation whole exome sequencing (NGS).

IVd. Anti-tumor immune response in peripheral blood, including serologic responses and analysis of T cell receptor (TCR) repertoires by deep sequencing.

IVe. Shift in quantitative laboratory peripheral blood parameters after the first 6 and 12 weeks of therapy.

OUTLINE: Patients are randomized to 1 of 2 treatment groups.

GROUP I:

INDUCTION: Patients receive nivolumab intravenously (IV) over 30 minutes every 2 weeks. Treatment repeats every 4 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive nivolumab IV over 30 minutes every 2 weeks. Treatment repeats every 4 weeks for up to 21 cycles in the absence of disease progression or unacceptable toxicity.

GROUP II:

INDUCTION: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 90 minutes. Treatment repeats every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive nivolumab IV over 30 minutes every 2 weeks. Treatment repeats every 4 weeks for up to 21 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 100 days, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal cancer with documented disease progression (disease not amendable to curative therapy); histologic confirmation of the original primary tumor is required via the pathology report; NOTE: patients with mucinous histology are NOT eligible; patients with carcinosarcoma histology are NOT eligible
* All patients must have measurable disease as defined by RECIST 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target" lesion to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Appropriate for study entry based on the following diagnostic workup:

  * History/physical examination within 28 days prior to registration
  * Imaging of target lesion(s) within 28 days prior to registration
  * Further protocol-specific assessments:

    * Recovery from effects of recent surgery, radiotherapy or chemotherapy
    * Free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
    * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
    * Any other prior therapy directed at the malignant tumor including chemotherapy, targeted agents, immunologic agents, and any investigational agents, must be discontinued at least 4 weeks prior to registration (6 weeks for nitrosoureas or mitomycin C)
    * Any prior radiation therapy must be completed at least 4 weeks prior to registration
    * At least 4 weeks must have elapsed since major surgery
* Patients are allowed to have received up to three prior cytotoxic regimens for treatment of their epithelial ovarian, fallopian tube, or primary peritoneal cancer; they must have had one prior platinum-based chemotherapeutic regimen for management of primary disease, possibly including intra-peritoneal therapy, consolidation, biologic/targeted (non-cytotoxic) agents or extended therapy (maintenance/consolidation) administered after surgical or non-surgical assessment; patients are allowed to have received, but are not required to have received, one to two cytotoxic regimens for management of recurrent or persistent disease; (for the purposes of this study poly adenosine diphosphate [ADP] ribose polymerase [PARP] inhibitors given for recurrent or progressive disease will be considered cytotoxic; PARP inhibitors given as maintenance therapy in continuation with management of primary disease will not be considered as a separate cytotoxic regimen); if two cytotoxic regimens had been received for management of recurrent or persistent disease, one of these regimens would have had to contain either a platinum or a taxane agent
* Performance status of 0, 1 or 2 within 28 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500/ul (within 14 days prior to registration)
* Platelets >= 100,000/ul (within 14 days prior to registration)
* Creatinine =< 1.5 x institutional/laboratory upper limit of normal (ULN) (within 14 days prior to registration)
* Bilirubin =< 1.5 x ULN; for patients with Gilbert's syndrome, bilirubin =< 3.0 mg/dL is acceptable (within 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (within 14 days prior to registration)
* Albumin >= 2.8 g/dL (within 14 days prior to registration)
* Adequate thyroid function within 28 days prior to registration defined as serum thyroid-stimulating hormone (TSH) in normal range
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* Platinum-free interval (PFI) - patients must have progressed < 12 months after completion of their last platinum-based chemotherapy; the date (platinum free interval) should be calculated from the last administered dose of platinum therapy to documentation of progression
* Adequate oxygen saturation via pulse oximeter within 28 days prior to registration (i.e., patient can NOT have CTCAE hypoxia grade 2 or greater)
* Left ventricular ejection fraction (LVEF) >= 50% (measured within 28 days of study entry)

Exclusion Criteria:

* Patients who have had prior therapy with nivolumab or with an anti-programmed cell death (PD)-1, anti-PD-ligand (L)1, anti-PD-L2, anti-cytotoxic T-lymphocyte-antigen (CTLA)-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune check point pathways
* History of severe hypersensitivity reaction to any monoclonal antibody
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies are excluded if there is any evidence of other malignancy being present within the last three years (2 years for breast cancer); patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy and radiotherapy for localized breast cancer, provided that it was completed more than 2 years prior to registration, and the patient remains free of recurrent or metastatic disease and hormonal therapy has been discontinued; patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis or thoracic cavity within the last three years are excluded; prior radiation for localized cancer of the head and neck or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients with uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure and unstable angina pectoris
* Patients with history of organ transplant
* Patients who are pregnant or nursing; women of child-bearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; WOCBP should use an adequate method to avoid pregnancy for 23 weeks after the last dose of investigational drug; WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IV/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab or nivolumab + ipilimumab; women must not be breastfeeding; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) do not require contraception; women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy and/or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 month amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level greater than 40 mIU/mL; if, following initiation of the investigational product(s), it is subsequently discovered that a study subject is pregnant or may have been pregnant at the time of investigational product exposure, including during at least 6 half-lives after product administration, the investigational product will be permanently discontinued in an appropriate manner (e.g., dose tapering if necessary for subject safety); the investigator must report this event and any outcomes by amendment through Cancer Therapy Evaluation Program (CTEP)-Adverse Event Reporting System (AERS); protocol-required procedures for study discontinuation and follow-up must be performed on the subject unless contraindicated by pregnancy (e.g., X-ray studies); other appropriate pregnancy follow-up procedures should be considered if indicated; in addition, the investigator must report and follow-up on information regarding the course of the pregnancy, including perinatal and neonatal outcome; infants should be followed for a minimum of 8 weeks
* History or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures which are not controlled with non-enzyme inducing anticonvulsants, any brain metastases and/or epidural disease, or history of cerebrovascular accident (cerebrovascular accident [CVA], stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months prior to the first date of study treatment
* In order for patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) to be eligible, they must be on a stable highly active antiretroviral therapy (HAART) regimen, have cluster of differentiation (CD)4 counts > 350, with no detectable viral load on quantitative polymerase chain reaction (PCR)
* Patients with treated hepatitis virus infections (hepatitis B or hepatitis C) are eligible if they have been definitively treated for 6 months, have no detectable viral load on quantitative PCR, and liver function tests (LFTs) meet eligibility requirements
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease, Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded; patient with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement (such as Hashimoto's thyroiditis), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Any of the following within 2 months of registration: active peptic ulcer disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, malabsorption syndrome; any of the following within 6 months of registration: intra-abdominal abscess, gastrointestinal obstruction requiring parenteral hydration and/or nutrition, gastrointestinal perforation; Note: complete resolution of an intra-abdominal abscess must be confirmed prior to registration even if the abscess occurred more than 6 months prior to registration
* No planned concomitant, non-protocol directed anti-cancer therapy
* Grade >= 2 peripheral neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2025-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitry Zamarin, Principal Investigator — NRG Oncology
Locations (201):
- United States (201):
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Sutter Davis Hospital, Davis, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Yale University, New Haven, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Emory Decatur Hospital, Decatur, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Rush-Copley Medical Center, Aurora, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Monongalia Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on 6/29/2015 and enrolled 49 patients. It temporarily closed on 10/7/2015 and awaited data maturation until 10/4/2016. The study reopened on 5/22/2017 and closed 8/28/2017 with a cumulative accrual of 100 patients
Groups:
- Treatment 1: Nivolumab: Nivolumab 3mg/kg IV once every 2 weeks x 4 doses (induction phase), followed by Nivolumab 3 mg/kg IV every 2 weeks (maintenance phase), for a maximum of 42 doses of maintenance therapy, until disease progression or until development of unacceptable toxicity, whichever comes first.
  1 Cycle = 4 weeks
- Treatment II: Nivolumab/Ipilimumab: Nivolumab 3mg/kg IV and Ipilimumab 1mg/kg IV once every 3 weeks x 4 doses (induction phase)*, followed by Nivolumab 3 mg/kg IV every 2 weeks (maintenance phase), for a maximum of 42 doses of maintenance therapy, until disease progression or until development of unacceptable toxicity, whichever comes first.
  1 Cycle = 3 weeks for induction phase
  1 Cycle = 4 weeks for maintenance phase
Period: Overall Study
Arm/Group | Treatment 1 | Treatment II
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment II | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Customized [Count of Participants; unit: Participants]
  18-49 years | 7 | 4 | 11
  50-59 ;years | 10 | 15 | 25
  60-69 years | 14 | 21 | 35
  >=70 years | 18 | 11 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 51 | 100
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 44 | 50 | 94
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 5 | 7
  White | 43 | 43 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: Complete and Partial Tumor Response by modified irRECIST. Per Response Evaluation Criteria In Solid Tumors Criteria (irRECIST) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Within 6 months of study entry
Population: All randomized patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 1 | Treatment II
Number analyzed (Participants) | 49 | 51
percentage of participants | 12.2 [5 to 23] | 31.4 [21 to 44]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time until disease progression, death, or date of last contact. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (irRECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: The duration of time from study entry to time of progression or death, whichever occurs first, an average of 3.9 months.
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment 1 | Treatment II
Number analyzed (Participants) | 49 | 51
months | 2.0 [1.9 to 2.7] | 3.9 [3.4 to 5.6]

3. Secondary Outcome: Duration of Overall Survival (OS)
Description: The observed length of life from randomization into the study to death or the date of last contact.
Time Frame: The duration of time from study entry to time of death or the date of last contact, assessed up to 5 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment 1 | Treatment II
Number analyzed (Participants) | 49 | 51
months | 21.8 [8.9 to NA] — Insufficient number of participants with events | 28.1 [12.6 to NA] — Insufficient number of participants with events

4. Secondary Outcome: Incidence of Adverse Events Grade 3 and Above
Description: Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 30 days after treatment ends
Population: All randomized patients.
Measure: Number; unit: number of adverse events
Arm/Group | Treatment 1 | Treatment II
Number analyzed (Participants) | 49 | 51
number of adverse events | 52 | 74

5. Other Pre Specified Outcome: Natural Anti-tumor Immunity in Tumor Infiltrating Lymphocytes and Tumor Cells
Description: Assessed with immunohistochemistry.
Time Frame: Baseline
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Markers of "Immunogenicity"
Description: Determined by the neo-epitope landscape using next-generation whole exome sequencing.
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Changes in Biomarkers
Description: Will assess the impact of biomarkers on tumor response, PFS, and OS.
Time Frame: Baseline to after the first 8 weeks of therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The average length of time adverse events were collected was 92 days.
Description: Eligible and treated participants were affected if they experienced grade 1-5 adverse event
Arm/Group | Treatment 1 | Treatment II
All-Cause Mortality (participants affected / at risk) | 24/49 | 21/51
Serious Adverse Events (participants affected / at risk) | 22/49 | 27/51
Other Adverse Events (participants affected / at risk) | 48/49 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=49) | Treatment II (N=51)
Cardiac Arrest (Cardiac disorders) | 1 | 0
Endocrine Disorders - Other (Endocrine disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Pain (General disorders) | 0 | 1
Edema Face (General disorders) | 0 | 1
Death Nos (General disorders) | 1 | 0
Infusion Related Reaction (General disorders) | 1 | 0
Hepatic Hemorrhage (Hepatobiliary disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 1
Infections And Infestations - Other (Infections and infestations) | 0 | 1
Serum Amylase Increased (Investigations) | 1 | 1
Platelet Count Decreased (Investigations) | 1 | 0
Lipase Increased (Investigations) | 0 | 4
Aspartate Aminotransferase Increased (Investigations) | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 | 0
Social Circumstances - Other (Social circumstances) | 1 | 0
Thromboembolic Event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=49) | Treatment II (N=51)
Hemolytic Uremic Syndrome (Blood and lymphatic system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 20 | 25
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 3 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 1 | 3
Chest Pain - Cardiac (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 2
Hearing Impaired (Ear and labyrinth disorders) | 2 | 2
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 2
Hypothyroidism (Endocrine disorders) | 2 | 11
Hyperthyroidism (Endocrine disorders) | 3 | 8
Watering Eyes (Eye disorders) | 0 | 1
Flashing Lights (Eye disorders) | 1 | 0
Eye Pain (Eye disorders) | 1 | 2
Glaucoma (Eye disorders) | 0 | 1
Blurred Vision (Eye disorders) | 5 | 7
Dry Eye (Eye disorders) | 0 | 5
Floaters (Eye disorders) | 1 | 1
Eyelid Function Disorder (Eye disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Dry Mouth (Gastrointestinal disorders) | 1 | 6
Colonic Stenosis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 19 | 24
Diarrhea (Gastrointestinal disorders) | 15 | 21
Vomiting (Gastrointestinal disorders) | 10 | 12
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 4 | 4
Stomach Pain (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 3
Abdominal Pain (Gastrointestinal disorders) | 16 | 21
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 3 | 3
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 25 | 27
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 7
Rectal Pain (Gastrointestinal disorders) | 0 | 1
Fecal Incontinence (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 4
Pain (General disorders) | 10 | 3
Neck Edema (General disorders) | 0 | 3
Malaise (General disorders) | 0 | 3
Irritability (General disorders) | 0 | 1
Flu Like Symptoms (General disorders) | 2 | 1
Non-Cardiac Chest Pain (General disorders) | 3 | 2
Edema Limbs (General disorders) | 5 | 12
Edema Face (General disorders) | 0 | 1
Fatigue (General disorders) | 32 | 38
Fever (General disorders) | 7 | 11
Gait Disturbance (General disorders) | 1 | 0
Chills (General disorders) | 3 | 2
Hypothermia (General disorders) | 0 | 1
Infusion Related Reaction (General disorders) | 1 | 1
Hepatic Hemorrhage (Hepatobiliary disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 2
Vaginal Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 1
Catheter Related Infection (Infections and infestations) | 1 | 0
Bronchial Infection (Infections and infestations) | 0 | 1
Bladder Infection (Infections and infestations) | 0 | 2
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 1
Radiation Recall Reaction (Dermatologic) (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Wound Complication (Injury, poisoning and procedural complications) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 0
Weight Loss (Investigations) | 5 | 7
Serum Amylase Increased (Investigations) | 5 | 8
Platelet Count Decreased (Investigations) | 7 | 7
Lymphocyte Count Decreased (Investigations) | 3 | 6
Lipase Increased (Investigations) | 9 | 7
Inr Increased (Investigations) | 2 | 3
Creatinine Increased (Investigations) | 7 | 10
Cholesterol High (Investigations) | 2 | 1
Neutrophil Count Decreased (Investigations) | 3 | 3
Carbon Monoxide Diffusing Capacity Decreased (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 1 | 3
White Blood Cell Decreased (Investigations) | 9 | 6
Aspartate Aminotransferase Increased (Investigations) | 19 | 16
Alkaline Phosphatase Increased (Investigations) | 10 | 7
Alanine Aminotransferase Increased (Investigations) | 14 | 11
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2 | 2
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 0
Hyponatremia (Metabolism and nutrition disorders) | 9 | 18
Hypomagnesemia (Metabolism and nutrition disorders) | 17 | 14
Hypokalemia (Metabolism and nutrition disorders) | 4 | 13
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 | 20
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 18 | 21
Hypercalcemia (Metabolism and nutrition disorders) | 5 | 4
Glucose Intolerance (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Anorexia (Metabolism and nutrition disorders) | 10 | 12
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 6
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 6 | 7
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 13
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Spasticity (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 0 | 1
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 19 | 19
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 3 | 0
Memory Impairment (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 0 | 2
Intracranial Hemorrhage (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 9 | 15
Facial Nerve Disorder (Nervous system disorders) | 0 | 1
Facial Muscle Weakness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Sinus Pain (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 7 | 7
Concentration Impairment (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Akathisia (Nervous system disorders) | 0 | 1
Libido Decreased (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 9
Depression (Psychiatric disorders) | 10 | 7
Confusion (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 8 | 5
Agitation (Psychiatric disorders) | 0 | 1
Urine Discoloration (Renal and urinary disorders) | 1 | 0
Urinary Urgency (Renal and urinary disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 2
Urinary Retention (Renal and urinary disorders) | 1 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 5
Urinary Tract Pain (Renal and urinary disorders) | 1 | 2
Urinary Frequency (Renal and urinary disorders) | 1 | 3
Proteinuria (Renal and urinary disorders) | 3 | 0
Hematuria (Renal and urinary disorders) | 2 | 3
Bladder Spasm (Renal and urinary disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 3
Vaginal Pain (Reproductive system and breast disorders) | 1 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 3
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 1
Perineal Pain (Reproductive system and breast disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 4
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 1
Dyspareunia (Reproductive system and breast disorders) | 2 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 19
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 15
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 7 | 19
Nail Discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 5
Thromboembolic Event (Vascular disorders) | 3 | 4
Hypotension (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 6 | 13
Hot Flashes (Vascular disorders) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT02498600/Prot_SAP_000.pdf